CLINICAL TRIAL: NCT05603689
Title: Effect of a Four-week Isocaloric Ketogenic Diet on Physical Performance at Very High Altitude: a Pilot Study
Brief Title: Effect of Isocaloric Ketogenic Diet on Physical Performance at High Altitude
Acronym: ICKD
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Clinique Romande de Readaptation (Network)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Single | Purpose: Basic Science
Other Study IDs: CRR
Record Dates: First submitted 2022-10-26; First posted 2022-11-03 (Actual); Last update posted 2022-11-03 (Actual); Status verified 2022-10

CONDITIONS: Ketogenic Dieting; Altitude Hypoxia; Physical Activity
MeSH Terms: conditions — Altitude Sickness; Motor Activity

STUDY DESIGN:
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Normal diet (Active Comparator): no limitations on food consumption.
  Interventions: Dietary Supplement: Isocaloric ketogenic diet
- Isocaloric ketogenic diet (Experimental): We defined ICKD as a daily CHOs ingestion < 30 to 50 g.d-1, without any limitation in fat consumption.
  Interventions: Dietary Supplement: Isocaloric ketogenic diet

INTERVENTIONS:
Dietary Supplement: Isocaloric ketogenic diet — The ICKD definition was based on the works of Sansone (2018) and Trimboli (2020). We defined ICKD as a daily CHOs ingestion < 30 to 50 g.d-1, without any limitation in fat consumption. Participants self-selected their own diet based on a list of advised and forbidden foods developed to fit the definition of ICKD. There were no instructions to limit calories.

SUMMARY:
A ketogenic diet (KD) reduces daily carbohydrates (CHOs) ingestion by replacing most calories with fat. KD is of increasing interest among athletes because it may increase their maximal oxygen uptake (VO2max), the principal performance limitation at high altitudes. The investigators examined the tolerance of a 4-week isocaloric KD (ICKD) under simulated hypoxia and the possibility of evaluating ICKD performance benefits with a maximal graded exercise bike test under hypoxia and collected data on the effect of the diet on performance markers and arterial blood gases.

DETAILED DESCRIPTION:
In a randomised single-blind cross-over model, 6 recreational mountaineers (age 24 to 44 years) will complete a 4-week ICKD followed or preceded by a 4-week habitual mixed western diet (HD). Performance parameters (VO2max, lactate threshold [LT], peak power [Ppeak]) and arterial blood gases (PaO2, PaCO2, pH, HCO3-) will be measured at baseline under two conditions (normoxia and hypoxia) as well as after a 4-week HD and 4-week ICKD under the hypoxic condition.

ELIGIBILITY:
Inclusion Criteria:

* Recreational mountaineers
* Familiarity with altitude (>2500 m above sea level) and males/females 20 to 45 years old.

Exclusion Criteria:

* high training load (such as professional athletes) or new planned training
* dietary restrictions.

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 8 (Actual)
Dates: Start 2020-09-01 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-09-23 (Actual)

PRIMARY OUTCOMES:
Performance test under hypoxic conditions | after 4 weeks of diet
  VO2max cycling test on ergometer

CONTACTS AND LOCATIONS:
Overall Officials: Lara Allet, PhD, Study Director — HESso
Locations (1):
- CRR, Sion, Switzerland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Chiarello N, Leger B, De Riedmatten M, Rossier MF, Vuistiner P, Duc M, Rapillard A, Allet L. Effect of a four-week isocaloric ketogenic diet on physical performance at very high-altitude: a pilot study. BMC Sports Sci Med Rehabil. 2023 Mar 20;15(1):37. doi: 10.1186/s13102-023-00649-9. PMID 36941621